CLINICAL TRIAL: NCT00272012
Title: Efficacy and Safety of Insulin Glulisine Given as a Single Injection at Breakfast + Insulin Glargine+OAD (Oral Antidiabetic Drug) vs Insulin Glulisine Given as a Single Injection at Main Meal+Insulin Glargine+OAD in Type 2 Diabetic Patients for Which Glycemic Control is Suboptimal Using Insulin Glargine+ OAD Alone
Brief Title: OPAL - Insulin Glulisine, Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Heinz Riederer / Medical Director, Sanofi-aventis Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR1964A_3507
Record Dates: First submitted 2006-01-02; First posted 2006-01-04 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin glulisine

INTERVENTIONS:
Drug: Insulin glulisine

SUMMARY:
Primary objective:

The primary study objective is to compare efficacy of Insulin glulisine, once a day at breakfast vs. Insulin glulisine given once a day at main meal in combination with insulin glargine + OAD in terms of change in HbA1c, from baseline to endpoint for the individual patient. The aim of the study is to demonstrate two-sided equivalence between the two therapy regimens receiving two different injection timing of Insulin glulisine.

Secondary objective:

Secondary study objectives are to compare efficacy and safety of Insulin glulisine, once a day at breakfast vs. Insulin glulisine given once a day at main meal in combination with insulin glargine + OAD in terms of:

* Change of fasting-, pre-/2h-postprandial-, mean daily and nocturnal blood glucose (baseline to endpoint)
* Change of fasting plasma glucose (baseline to endpoint)
* Response rate: Responders will be those patients with HbA1c smaller than 7.0% at study endpoint
* Insulin dose (rapid-acting, basal and total daily doses)
* Weight, body-mass index
* Hypoglycemic events
* Adverse events

ELIGIBILITY:
Inclusion criteria:

* Type 2 Diabetes mellitus, previously treated with combination therapy of insulin glargine + OAD (maximal tolerated dose / approved in combination with insulin according to local SPCs (Summary of Product Characteristics), not including use of a-glucosidase inhibitors) for at least 3 months
* Pre-screening HbA1c value greater/equal 7% - smaller/equal 9%
* FBG (Fasting Blood Glucose) smaller/equal 120 mg/dl (6.6 mmol/l)
* Women are either not of childbearing potential (surgically sterile, or postmenopausal for more than 2 years) or are not pregnant and agree to use a reliable contraceptive measure for the duration of the study. Reliable contraceptive measures include the following: systemic contraceptive (oral, implant, injections), diaphragm with intravaginal spermicide, cervical cap, intrauterine device, or condom with spermicide.
* Ability and willingness to perform blood glucose monitoring using the sponsor-provided blood glucose meter and subject diary at home

Exclusion criteria:

* More than two FBG greater 120 mg/dl (6.6 mmol/l) as measured on 5 consecutive days before visit II
* Active proliferative diabetic retinopathy, as defined by the application of focal or panretinal photocoagulation or vitrectomy, in the 6 months prior to visit 1, or any other unstable (rapidly progressing) retinopathy that may require surgical treatment (including laser photocoagulation)
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult
* Known impaired hepatic and renal function
* History of drug or alcohol abuse
* History of hypersensitivity to insulin or insulin analogues or any of the excipients in the Insulin glulisine formulation
* Treatment with any investigational drug in the last month before visit I
* Pregnant or breast-feeding women, or women planning to become pregnant during the study
* Treatment or likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Night shift workers if they are unable to comply with the treatment regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2004-07; Primary Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c. | from baseline to study endpoint.

SECONDARY OUTCOMES:
Change of pre-, 2 h postprandial and nocturnal blood glucose values | 8-point profile
Fasting blood glucose | 8-point blood glucose profile values
Responder rate HbA1c smaller 7 % | at study endpoint
Insulin dose | rapid-acting, basal and total daily doses
Weight, BMI | study follow-up
Hypoglycemic events | study follow-up
Adverse events. | study follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Landgraf, Dr., Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Berlin, Germany